CLINICAL TRIAL: NCT07396870
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dosed Phase II Clinical Study to Evaluate the Efficacy and Safety of LPM787000048 Maleate Extended-Release Tablets (LY03020) in Acutely Psychotic Adult Subjects With Schizophrenia
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of LY03020 in Acutely Psychotic Participants With Schizophrenia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03020/CT-CHN-204
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03020 (Experimental): Subjects will take LY03020 from Day 1 to Day 48
  Interventions: Drug: LY03020
- Placebo (Placebo Comparator): Subjects will take Placebo from Day 1 to Day 48
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03020 — administered orally
  Arms: LY03020
Drug: Placebo — administered orally
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled, fixed-dosed phase II clinical study to evaluate the efficacy and safety of LY03020 in chinese acutely psychotic adult subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and their guardians sign informed consent voluntarily.
* Male or female subject aged 18 to 65 years (inclusive).
* Subject meets DSM-5 criteria for schizophrenia and confirmed using the Mandarin for China Translation Version 7.0.2).
* According to the investigator's assessment, subject has an acute exacerbation or relapse of schizophrenia requiring hospitalization (no longer than 2 months). Continuing hospitalization does not exceed 2 weeks for patients with acute psychotic exacerbation or relapse that require the hospitalization prior to screening.
* Subject must have a PANSS total score ≥ 80 and a PANSS item score ≥ 4 (moderate) on 2 or more of the following PANSS items: delusions(P1), conceptual disorganization(P2), hallucinations(P3), and suspicion, victimization (P6) at screening and baseline.
* Subject must have a CGI-S score ≥ 4 at screening and baseline.

Exclusion Criteria:

* - Subject who has a history or presence of symptoms consistent with a major psychiatric disorder other than schizophrenia as defined by DSM-5;
* According to the investigator's assessment, subject has a treatment-resistant schizophrenia;
* Subject who has a history or presence of symptoms consistent with neuroleptic malignant syndrome (NMS);
* Subject has received electroconvulsive therapy treatment within 3 months prior to screening or is expected to require ECT during the study;
* History of suicide attempts (including actual attempts, interrupted attempts, or failed attempts) within 1 year prior to screening or suicidal ideation within 6 months prior to screening, defined as affirmative responses ("yes") to question 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening/baseline;
* History or presence of the following treatments:

Within 1 week prior to randomization or within 5 half lives (whichever is longer), subject has been treated with short acting antipsychotic drugs or other psychoactive drugs (such as antidepressants, mood stabilizers, and antiepileptic drugs), except for anti-anxiety drugs or sedative hypnotic drugs that can be used according to the protocol; Within two treatment cycles prior to randomization, subject has used long-acting antipsychotic drugs; Within 4 weeks prior to randomization, subject has used monoamine oxidase inhibitors (MAOIs); Previously used sufficient amounts and periods of clozapine for the treatment of schizophrenia;

* Congenital long QT syndrome; uncontrolled or severe cardiovascular disease, including NYHA class II or higher congestive heart failure, unstable angina, myocardial infarction within 6 months prior to screening, or presence of treatment-requiring severe arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) at screening; resting heart rate <50 beats per minute (bpm) and the abnormality has clinical significance according to the researchers' assessment at screening/baseline; or QTc >450 ms (male) / QTc >460 ms (female) based on Fridericia's formula-corrected measurements and the abnormality has clinical significance according to the researchers' assessment at screening/baseline;
* Subjects experienced a history of keratopathy, fundus disease, increased intraocular pressure, or angle-closure glaucoma;.
* Subjects with a history of orthostatic hypotension or syncope.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Positive and Negative Syndrome Scale (PANSS) total score | baseline to week 6 of maintenance treatment
  The total score is 30-210, higher score is indicative of greater symptomatology.

SECONDARY OUTCOMES:
Change from Baseline in PANSS Positive subscale score | baseline to week 6 of maintenance treatment
  The PANSS Positive subscale score is 7-49, higher score is indicative of greater symptomatology.
Change from Baseline in PANSS Negative subscale score | baseline to week 6 of maintenance treatment
  The PANSS Negative subscale score is 7-49, higher score is indicative of greater symptomatology.
Change from Baseline in PANSS General Psychopathology subscale score | baseline to week 6 of maintenance treatment
  The PANSS General Psychopathology subscale score is 16-112, higher score is indicative of greater symptomatology.
Change from Baseline in Clinical Global Impression-Severity (CGI-S) score | baseline to week 6 of maintenance treatment
  CGI-S is 0-7 with higher score is indicative of greater symptomatology
The Incidence of Overall AEs | baseline to week 6 of maintenance treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing AnDing Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No